CLINICAL TRIAL: NCT05968196
Title: Clinicopathological Characteristics of Hürthle Cell Carcinoma and Follicular Thyroid Carcinoma Without Completion Thyroidectomy
Brief Title: Hürthle Cell Carcinoma and Follicular Thyroid Carcinoma
Acronym: HCC and FTC
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kwangsoon Kim, Assistant Professor, The Catholic University of Korea
Other Study IDs: noar99
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Huerthle Cell Carcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FTC: Follicular thyroid carcinoma
- HCC: Hurthle cell carcinoma

SUMMARY:
The goal of this retrospective study is to evaluate in patients with HCC and FTC who underwent lobectomy. The main questions it aims to answer are:

* The necessity of completion thyroidectomy based on the clinicopathological characteristics
* Prognosis Participants underwent thyroid lobectomy Researchers compared HCC and FTC groups to see the prognosis after lobectomy.

DETAILED DESCRIPTION:
Background The prognosis of Hürthle cell carcinoma (HCC) and follicular thyroid carcinoma (FTC) is poorly understood. These types of cancers are usually confirmed after diagnostic lobectomy. We aimed to evaluate the clinicopathological characteristics and prognoses of patients with HCC and FTC who did not undergo completion thyroidectomy.

Materials and Methods We screened 221 patients diagnosed with FTC or HCC after thyroid lobectomy at Yonsei Severance Hospital between January 2000 and December 2020. After excluding patients who underwent complete thyroidectomy, 184 patients with FTC and 37 patients with HCC were included.

ELIGIBILITY:
Inclusion Criteria:

* Follicular thyroid carcinoma
* Hurthle cell carcinoma
* Lobectomy

Exclusion Criteria:

* Completion thyroidectomy
* Total thyroidectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in FTC and HCC who underwent thyroid lobectomy
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From January 2000 to March 2023
  a comparison of disease-free survival (DFS) between FTC and HCC groups

SECONDARY OUTCOMES:
TNM stage | From January 2000 to March 2023
  a comparison of TNM stage between FTC and HCC groups

IPD SHARING:
Plan to Share IPD: Undecided